CLINICAL TRIAL: NCT02867124
Title: Long-acting Naltrexone for Pre-release Prisoners: A Randomized Trial of Mobile Treatment
Brief Title: Long-acting Naltrexone for Pre-release Prisoners
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FriendsResearch; R01DA040636 (NIH)
Record Dates: First submitted 2016-08-08; First posted 2016-08-15 (Estimated); Last update posted 2026-02-03 (Actual); Status verified 2024-02

CONDITIONS: Opiate Addiction
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Residence Characteristics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vivitrol at place of residence (Experimental): One injection of long-acting naltrexone (XR-NTX) in prison, followed by 6 monthly injections post-release at the participants's place of residence utilizing mobile medical treatment
  Interventions: Drug: XR-NTX; Other: place of residence
- Vivitrol at opioid treatment program (Active Comparator): One injection of long-acting naltrexone (XR-NTX) in prison, followed by 6 monthly injections post-release at a community opioid treatment program.
  Interventions: Drug: XR-NTX; Other: opioid treatment program

INTERVENTIONS:
Drug: XR-NTX — Vivitrol
  Other Names: long-acting naltrexone
Other: place of residence — One injection of XR-NTX in prison, followed by 6 monthly injections post-release at place of residence
  Other Names: residence
  Arms: Vivitrol at place of residence
Other: opioid treatment program — One injection of XR-NTX in prison, followed by 6 monthly injections post-release at a community opioid treatment program
  Other Names: OTP
  Arms: Vivitrol at opioid treatment program

SUMMARY:
This proposed five-year study will focus on whether the addition of providing XR-NTX treatment at a patients' place of residence will increase adherence and thus efficacy of the medication.Following initial screening, informed consent, and medical examination, pre-release prisoners at each facility will be block randomized (N=240) within gender to either: Condition 1. XR-NTX-OTx (n=120): One injection of XR-NTX in prison, followed by six monthly injections post-release in the community at an opioid treatment program; or Condition 2. XR-NTX+MMTx (n=120): One injection of XR-NTX in prison, followed by six monthly injections post-release in the community at the patient's place of residence.

DETAILED DESCRIPTION:
Disorders involving opioid use are a severe problem among jail and prison inmates. Inmates in the US, Canada, Australia, and many European and Asian nations have disproportionately higher rates of opioid use disorders than their general populations. Scarce resources are provided for corrections-based substance use treatment in many nations, and many inmates with OUDs remain untreated. The use of long-acting, injectable naltrexone (XR-NTX) may be a promising form of treatment for pre-release prisoners. Naltrexone blocks the intoxicating and reinforcing effects of opioids, but has no opioid-like effects. This proposed five-year study will focus on whether the addition of providing XR-NTX treatment at a patients' place of residence will increase adherence and thus efficacy of the medication. Project implementation will occur at five pre-release prisons under the jurisdiction of the Maryland Department of Public Safety and Correctional Services (MDPSCS): 1) Metropolitan Transition Center (MTC) for men; 2) Baltimore Pre-Release Unit (BPRU) for men; 3) Jessup Pre-Release Unit (JPRU) for men; 4) Baltimore City Correctional Center (BCCC) and 5) Maryland Correctional Institution (MCI) for Women. Following initial screening, informed consent, and medical examination, pre-release prisoners at each facility will be block randomized (N=240) within gender to either: Condition 1. XR-NTX-OTx (n=120): One injection of XR-NTX in prison, followed by six monthly injections post-release in the community at an opioid treatment program; or Condition 2. XR-NTX+MMTx (n=120): One injection of XR-NTX in prison, followed by six monthly injections post-release in the community at the patient's place of residence. All participants will be confirmed opiate-free by urine test and negative naloxone and oral naltrexone tests, and evaluated monthly for seven months and 12 months after release from prison. The proposed study has two specific aims: Aim1. To compare the two study conditions in terms of: a) XR-NTX treatment adherence; b) opioid use; c) criminal activity; d) re-arrest; e) re-incarceration; and f) HIV risk-behaviors (i. needle use; ii. risky sexual behaviors). Aim 2. To determine if the number of months of post-release XR-NTX treatment is related to outcome (a-f above), and if so, is there a point at which XR-NTX v. Non-XR-NTX equilibrates? This would help determine the number of injections, important because of XR-NTX cost. Many individuals in the criminal justice system drop out of treatment and therefore increasing ways to improve adherence by attempting to: 1) expand capacity; and 2) implement access by providing treatment at their place of residence may positively impact outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female inmate at MTC, BPRU, JPRU, BCCC, or MCIW and be eligible for release within 30 days
* History of opiate disorder [meeting DSM-V criteria of dependence at the time of incarceration]
* Suitability for XR-NTX treatment as determined by medical evaluation
* Currently opioid-free by history, with negative urine for all opioids and no signs of opiate withdrawal
* Willingness to enroll in XR-NTX treatment in prison [not currently in or planning to pursue agonist (methadone, buprenorphine) treatment at release]
* Planning to live in Baltimore City or County.
* Inmates not meeting the opioid-dependence criterion will be eligible if they were treated in an opioid agonist treatment program during the year before incarceration

Exclusion Criteria:

* Liver function test levels greater than three times normal
* Active medical illness that may make participation hazardous (e.g., unstable diabetes, heart disease). Adequately treated medical conditions are acceptable
* Untreated psychiatric disorder that may make participation hazardous (e.g., untreated psychosis, bipolar disorder with mania). Adequately treated psychiatric disorders and appropriate psychotropic medications will be allowed
* History of allergic reaction to XR-NTX
* Current chronic pain diagnosis for which opioids are prescribed
* Creatinine above normal limits
* Pregnancy (for women)
* Breast-feeding (for women)
* Suicidal ideation (within the past 6-months)
* Body Mass Index (BMI) > 40
* Unadjudicated charges that may result in transfer to another facility and/or additional prison time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
treatment adherence | six months
  XR-NTX+ MMTx vs. XR-NTX-OTx following release from prison
Any illicit opioid used | 1,2,3,4,5,6,7 and 12-months following release from prison
  defined as continuous counts of days and urine toxicologies for heroin or other illicit opioid
re-arrest | 12-months following release from prison
  Re-arrest will be assessed using self-report on the Arrests and Days Incarcerated form and from Official Records received from the Maryland Department of Public Safety and Correctional Services
re-incarceration | 12-months following release from prison
  Re-incarceration will be assessed using self-report on the Arrests and Days Incarcerated form and from Official Records received from the Maryland Department of Public Safety and Correctional Services
criminal activity | 1,2,3,4,5,6,7 and 12-months following release from prison
  Self-reported crime days will be defined as continuous counts of days collected from the Addiction Severity Index and Time Line Follow-Back
Injection drug use and HIV sexual risk factors | 6 and 12-months following release from prison
  Injection drug use and HIV sexual risk factors will be measured using the Risk Assessment Battery.

SECONDARY OUTCOMES:
Treatment Group Equilibration | 6 and 12-months following release from prison
  time point at which the trajectories for use in the two treatment groups cross

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Gordon, DPA, Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Maryland Department of Public Safety and Correctional Services, Towson, Maryland, United States

REFERENCES:
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086
- [Derived] Gordon MS, Vocci FJ, Fitzgerald TT, O'Grady KE, O'Brien CP. Extended-release naltrexone for pre-release prisoners: A randomized trial of medical mobile treatment. Contemp Clin Trials. 2017 Feb;53:130-136. doi: 10.1016/j.cct.2016.12.015. Epub 2016 Dec 20. PMID 28011389

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT02867124/Prot_SAP_000.pdf